CLINICAL TRIAL: NCT06242275
Title: Perioperative Salivary Alpha-amylase as a Predictor of Delirium After Lower Extremity Vascular Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ِAhmed Mohamed Ibrahim, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Other Study IDs: 36264PR462/12/23
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Salivary Alpha-amylase; Delirium; Lower Extremity; Vascular Bypass Surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative delirium (POD) group: Patients who will develop postoperative delirium
  Interventions: Diagnostic Test: Salivary Alpha-amylase
- No Postoperative delirium (POD) group: Patients who will not develop postoperative delirium
  Interventions: Diagnostic Test: Salivary Alpha-amylase

INTERVENTIONS:
Diagnostic Test: Salivary Alpha-amylase — Saliva samples will be obtained using a saliva collection system and salivary Alpha-amylase (SAA) level will be measured preoperatively, immediately postoperative, at the end of the 1st, 2nd, and 3rd postoperative days. For sampling, the swab will be placed into the patient's mouth for 2-5min by a specially trained nurse.
  A minimum of 0.2mL of saliva will be needed as per the manufacturer's recommendations to saturate the swab.

SUMMARY:
The aim of this study is to evaluate the role of salivary Alpha-amylase as a predictor biomarker of POD in elderly patients undergoing limb bypass surgery.

DETAILED DESCRIPTION:
Delirium is a neuropsychiatric syndrome that is characterized by the sudden onset of altered awareness, decreased ability to maintain attention, and disorders of the mental process. The pathophysiology of Postoperative delirium (POD) is related to postoperative neuroinflammation.

Biomarkers not only indicate a certain pathological state, but also provide information about disease activity and progression. Although several biomarkers are reported to predict POD, biomarkers with high sensitivity and specificity are still lacking.

Biochemical parameters associated with complement cascade (C3a, C3, C5a) and inflammatory response (IL-17A, IL-33, E-selectin, MMP9) were involved in neurocognitive regulation.

Salivary alpha amylase (SAA) enzyme is one of the most important enzyme compositions in the saliva that accounts for 40% to 50% of the total salivary proteins, and most of it is secreted from the parotid gland. SAA is locally produced by the highly differentiated epithelial acinar cells of the exocrine salivary glands, mostly of the parotid glands and plays an important role in carbohydrate hydrolysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status III.
* Undergoing lower extremity vascular surgery under general anesthesia.

Exclusion Criteria:

* Patients who used any medication that could affect salivary glands (such as antihypertensive, antidepressants or antipsychotic drugs).
* Inability to communicate.
* History of psychiatric diseases or previous stroke
* Previous history of pod.
* Those with smoking and drinking habits.
* Pregnant female.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 60 patients aged ≥ 65 years, both sexes, American Society of Anesthesiologists (ASA) physical status III, undergoing lower extremity vascular surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
The accuracy of salivary alpha-amylase as a predictor of postoperative delirium | 3rd day postoperatively
  The accuracy of salivary alpha-amylase will be measured by saliva samples which will be obtained using a saliva collection system and SAA level will be measured preoperatively, immediately postoperative, at the end of the 1st, 2nd, and 3rd postoperative days.

SECONDARY OUTCOMES:
Incidence of postoperative delirium | first 5 days after surgery
  Incidence of postoperative delirium will be measured.
Correlation of salivary alpha-amylase with C-reactive protein | 24 hours postoperatively
  Correlation of salivary alpha-amylase with C-reactive protein will be assessed.
Correlation of salivary alpha-amylase with average pain score | 24 hours postoperatively
  Correlation of salivary alpha-amylase with average pain score will be assessed. Pain score will be assessed using numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable.
Correlation of salivary alpha-amylase with morphine consumption | 24 hours postoperatively
  Correlation of salivary alpha-amylase with morphine consumption will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.